CLINICAL TRIAL: NCT05674357
Title: Training in Evidence-based Treatments in Psycho-Oncology
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Jamie Jacobs, Principal Investigator, Massachusetts General Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 22-517
Record Dates: First submitted 2022-12-21; First posted 2023-01-06 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2025-12

CONDITIONS: Distress, Emotional; Depression, Anxiety; Fatigue; Pain; Insomnia
Keywords: CBT; Cognitive-Behavioral Therapies; Emotional Distress; Anxiety; Depression; Symptom-Related Distress
MeSH Terms: conditions — Depression; Anxiety Disorders; Fatigue; Pain; Sleep Initiation and Maintenance Disorders | interventions — Caregivers

STUDY DESIGN:
Intervention Model Description: There will be two groups in this study- one is patient and caregiver participants (n=100) and the other is therapist participants (n=15). Therapist participants will deliver evidence-based therapy treatments to patients participants. Outcomes in each group will not be compared to each other.
Masking Description: There will be two groups in this study- one is patient and caregiver participants (n=100) and the other is therapist participants (n=15). Therapist participants will deliver evidence-based therapy treatments to patients participants. Outcomes in each group will not be compared to each other.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Individualized Evidence-Based Therapy in Cancer (Patients and Caregivers) (Experimental): This arm will enroll patient and caregiver participants receiving evidence-based therapy as part of the protocol.
  Participants will complete:
  * 6-16 sessions of therapy 1x/week. Sessions are virtual or in-person at the Massachusetts General Hospital Cancer Center.
  * Surveys and questionnaires pre- and post-treatment.
  At the discretion of the therapist and the supervising therapist, the participant may receive up to 4 booster sessions after completion of the specific treatment protocol.
  Interventions: Behavioral: Individualized Evidence-Based Therapy in Cancer (Patients and Caregivers)
- Training in Individualized Evidence-Based Therapy in Cancer (Therapists) (Experimental): This arm will enroll therapist participants as part of the protocol. Therapists participants will enroll in the study and receive training in delivering evidence-based therapy to patients in the cancer center. Therapists will complete pre and post-measures of therapist self-efficacy and competence, as well as a semi-structured exit interview.
  Interventions: Behavioral: Training in Individualized Evidence-Based Therapy in Cancer (Therapists)

INTERVENTIONS:
Behavioral: Individualized Evidence-Based Therapy in Cancer (Patients and Caregivers) — The intervention will mirror clinical care in psycho-oncology in which the therapist, collaboratively with their supervisor, will choose specific components of the following evidence-based treatments to administer based on the clinical presentation of the patient or caregiver and referring problem.
  * Cognitive Behavioral Therapy (CBT)
  * Acceptance Commitment Therapy (ACT)
  * Mindfulness-Based Cognitive Therapy (MBCT)
  * Mindfulness-Based Stress Reduction (MBSR)
  * Meaning-Centered Psychotherapy (MCP)
  * Cognitive Behavioral Therapy for Insomnia (CBT-I)
  * CBT for pain
  * CBT for fatigue
  * CBT for nausea
  Arms: Individualized Evidence-Based Therapy in Cancer (Patients and Caregivers)
Behavioral: Training in Individualized Evidence-Based Therapy in Cancer (Therapists) — Enrolled therapist participants will receive training in evidence-based therapies and deliver therapy to patient and caregiver participants.
  Arms: Training in Individualized Evidence-Based Therapy in Cancer (Therapists)

SUMMARY:
The goal of this research study is to train psychotherapists to administer individualized evidence-based psychotherapies in a cancer care setting to patients and caregivers with elevated levels of distress.

The intervention will mirror clinical care in psycho-oncology in which the therapist, collaboratively with their supervisor, will choose specific components of the following evidence-based treatments to administer based on the clinical presentation of the patient or caregiver and referring problem.

* Cognitive Behavioral Therapy (CBT)
* Acceptance Commitment Therapy (ACT)
* Mindfulness-Based Cognitive Therapy (MBCT)
* Mindfulness-Based Stress Reduction (MBSR)
* Meaning-Centered Psychotherapy (MCP)
* Cognitive Behavioral Therapy for Insomnia (CBT-I)
* CBT for other cancer-related physical symptoms like pain, fatigue, and nausea.

Participation in this research study is expected to last about 26 weeks.

It is expected that about 75 patients, 25 caregivers, and 15 therapists will take part in this research study.

DETAILED DESCRIPTION:
This is a single-arm, behavioral intervention study to train psychotherapists to administer individualized evidence-based psychotherapies in a cancer care setting to patients and caregivers with elevated levels of distress related to their illness, treatment and/or caregiving responsibilities. For participants with cancer and their caregivers, common treatment goals include improving health behaviors, reducing psychological symptoms that may exacerbate medical disability, and/or improving functional status.

Research procedures include screening for eligibility, completion of surveys and questionnaires, and virtual or in-person therapy sessions.

The intervention will mirror clinical care in psycho-oncology in which the therapist, collaboratively with their supervisor, will choose specific components of the following evidence-based treatments to administer based on the clinical presentation of the patient or caregiver and referring problem.

* Cognitive Behavioral Therapy (CBT)
* Acceptance Commitment Therapy (ACT)
* Mindfulness-Based Cognitive Therapy (MBCT)
* Mindfulness-Based Stress Reduction (MBSR)
* Meaning-Centered Psychotherapy (MCP)
* Cognitive Behavioral Therapy for Insomnia (CBT-I)
* CBT for other cancer-related physical symptoms like pain, fatigue, and nausea.

Participation in this research study is expected to last about 26 weeks.

It is expected that about 75 patients, 25 caregivers, and 15 therapists will take part in this research study.

Patient or caregiver participants will be those who a) are currently receiving oncology care, including active treatment and/or surveillance, or caring for someone currently receiving oncology care, b) report elevated levels of distress (≥ 3 on the NCCN Distress Thermometer), c) report that their distress or presenting concerns are related to their illness, their treatment(s), and/or their caregiving experience and d) have a clinical presentation that matches an evidence-based treatment (e.g., CBT-I for insomnia/sleep disturbance) for cancer-related distress per the therapist and the supervising therapist's discretion. The investigators aim to recruit up to 75 patient and 25 caregiver participants to this study over the course of 5 years. Therapist participants will be fellows or residents in the Mass General's Center for Psychiatric Oncology & Behavioral Sciences. The investigators aim to include up to 15 therapist participants over the course of this 5-year study. The study period for therapist participation would be up to 3 years, and would end either at a) 3 years, b) the point at which the therapist obtains licensure and transitions to faculty member, c) the time the therapist leaves MGH.

ELIGIBILITY:
Patient Inclusion Criteria:

* Adults > 18 years of age.
* Currently receiving oncology treatment/care at the MGH Cancer Center, including active treatment and/or surveillance.
* Reports elevated levels of distress on the National Comprehensive Cancer Network (NCCN) Distress Thermometer > 3.
* Reports distress or presenting problem is related to patients' illness and/or treatment (e.g., cancer treatment).
* Has a clinical presentation that matches an evidence-based treatment (e.g., CBT-I for insomnia/sleep disturbance) for cancer-related distress per therapist and supervising therapist discretion.
* Located in the state of Massachusetts for the duration of sessions.

Caregiver Inclusion criteria:

* Adults > 18 years of age
* Currently caring for someone receiving oncology treatment/care at the MGH Cancer Center, including active treatment and/or surveillance
* Reports elevated levels of distress on the National Comprehensive Cancer Network (NCCN) Distress Thermometer > 3
* Reports distress or presenting problem is related to caregiving
* Has a clinical presentation that matches an evidence-based treatment (e.g., CBT-I for insomnia/sleep disturbance) for caregiving-related distress per therapist and supervising therapist discretion
* Located in the state of Massachusetts for the duration of sessions

Patient Exclusion Criteria:

* Has uncontrolled psychosis, active suicidal ideation, or psychiatric hospitalization within the past year (assessed through EHR review and screening session using the QuickSCID-5), indicating the need for tailored treatment referral to specialty mental healthcare outside of psycho-oncology or to a higher level of care such as an intensive outpatient program (IOP).
* Has a cognitive impairment that prohibits participation in the study (assessed through EHR review and screening session).
* Currently participating in group or individual evidence-based psychotherapy treatment or other psychosocial intervention trial.
* Has an alcohol or substance dependence (other than nicotine dependence) in the past 8 weeks (assessed through EHR review and screening session using the QuickSCID-5), indicating the need for tailored treatment referral to specialty mental healthcare outside of psycho-oncology or to a higher level of care such as an intensive outpatient program (IOP).

Therapist Inclusion criteria:

-Current appointment as a clinical psychology fellow or psychiatry resident at the Massachusetts General Hospital or equivalent designation.

Therapist Exclusion criteria:

-Obtained licensure as a clinical psychologist in any state.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 115 (Estimated)
Dates: Start 2023-01-09 (Actual); Primary Completion 2028-01-01 (Estimated); Study Completion 2029-01-01 (Estimated)

PRIMARY OUTCOMES:
Evidence-Based Treatment Acceptability | up to 26 weeks
  Patients and caregivers will report acceptability of evidence-based treatment delivered by therapists receiving training in psycho-oncology on the Client Satisfaction Questionnaire (acceptability criteria: >75% of patients score ≥ the CSQ's midpoint [3]).
  Defined by the Client Satisfaction Questionnaire (CSQ), a 3-item, validated measure to assess satisfaction with services provided to the participant. Each item is answered on a scale of 1-4 with a total score range of 3-12. Acceptability criteria is > 75% of participants with a score ≥ the CSQ's midpoint.

SECONDARY OUTCOMES:
Coping Self-Efficacy | up to 26 weeks
  Defined by the Measures of Current Status Part A (MOCS-A), a 13-item scale which measures participants' current self-perceived ability on several skills. Each of the 13 items is answered on a scale of 0 (I cannot do this at all) to 4 (I can do this extremely well).
Patient Quality of Life (FACT-G) | up to 26 weeks
  Defined by the Functional Assessment of Cancer Therapy General (FACT-G), a 27-item questionnaire designed to measure four domains of health-related QOL in cancer participants. Items are rated on 5-item Likert scale.
Caregiver Quality of Life (CarGOQoL) | up to 26 weeks
  Defined by the CareGiver Quality of Life Questionnaire (CarGOQoL), a 29-item questionnaire designed to measure ten dimensions of caregivers of patients with cancer's QOL. Items are rated on a 5-item Likert scale.

CONTACTS AND LOCATIONS:
Overall Officials: Jamie Jacobs, Ph.D, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital Cancer Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
The Dana-Farber / Harvard Cancer Center encourages and supports the responsible and ethical sharing of data from clinical trials. De-identified participant data from the final research dataset used in the published manuscript may only be shared under the terms of a Data Use Agreement. Requests may be directed to: [contact information for Sponsor Investigator or designee]. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP
Time Frame: Data can be shared no earlier than 1 year following the date of publication.
Access Criteria: Contact the Partners Innovations team at http://www.partners.org/innovation